CLINICAL TRIAL: NCT07338136
Title: Computer Guided Split Thickness Versus Full Thickness Flap Buccal Bone Lid Approach in Hard Mandibular Pathosis: Randomized Control Trial RCT
Brief Title: Computer Guided Split Thickness Versus Full Thickness Flap Buccal Bone Lid Approach in Hard Mandibular Pathosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Salah Azab, doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: omfs3-3-6
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Mandibular Diseases; Guided Surgery; Guided Surgery Accuracy
Keywords: buccal bone lid; split thickness flap; computer guided surgery; mandibular pathosis; impacted tooth
MeSH Terms: conditions — Mandibular Diseases; Tooth, Impacted

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer guided full thickness flap for buccal bone lid approuch in hard mandibular pathosis (Active Comparator): * After anaesthesia administration, a full-thickness flap will be elevated with one or two releasing incisions.
  * Guide will be seated according to the pre-planned position.
  * The bone lid osteotomies will be prepared following the internal profile of the guide using a piezoelectrical device.
  * The guide will be removed, and the bone lid will be completed and detached.
  * The bony lid will be saved in saline solution until fixation.
  * Pathosis will be removed completely, and the lid will be returned and fixed to its original position using one or more screw.
  * Suturing with primary closure will be obtained.
  * Immediate post-operative CBCT will be taken
  Interventions: Procedure: computer guided split thickness flap for buccal bone lid approuch
- computer guided split thickness flap for buccal bone lid approuch in hard mandibular pathosis (Experimental): * After anesthesia administration, a split-thickness flap will be elevated.
  * Guide will be seated according to the pre-planned position.
  * Periosteal incision will be performed following the external profile of the surgical guide.
  * The guide will be removed, and a minimum periosteal reflection will be done.
  * The guide will be placed again, and the bone lid osteotomies will be prepared following the internal profile of the guide using piezoelectrical device.
  * The guide will be removed again, and the bone lid will be completed and detached with its attached periosteum.
  * The bony lid with its attached periosteum will be saved in saline solution until fixation.
  * Pathosis will be removed completely, and the lid will be returned and fixed to its original position using one or more screw.
  * Suturing with primary closure will be obtained.
  Interventions: Procedure: computer guided split thickness flap for buccal bone lid approuch

INTERVENTIONS:
Procedure: computer guided split thickness flap for buccal bone lid approuch — * After anesthesia administration, a split thickness flap will be elevated.
  * Guide will be seated according to the pre-planned position.
  * Periosteal incision will be performed following the external profile of the surgical guide.
  * The guide will be removed and minimum periosteal reflection will be done.
  * The guide will be placed again and the bone lid osteotomies will be prepared following the internal profile of the guide using piezoelectrical device.
  * The guide will be removed again, and the bone lid will be completed and detached with its attached periosteum.
  * The bony lid with its attached periosteum will be saved in saline solution until fixation.
  * Pathosis will be removed completely, and the lid will be returned and fixed to its original position using one or more screw.
  * Suturing with primary closure will be obtained.
  * Immediate post-operative CBCT will be taken

SUMMARY:
* Full thickness Buccal bone lid approach is well known and well reported technique with a superiority on preserving bone volume and better bone healing especially when done using piezoelectrical devices when compared to conventional technique for management of mandibular pathosis, however periosteum disturbance have a negative role regarding vascularity and bone healing, by comparing the split thickness VS full thickness flap design with buccal bone lid approach, this study will highlight if the periosteum preserved attached to the lid improve the healing on mandibular bony pathosis.
* Aim of the study:

determine the effect of split thickness flap vs full thickness flap using a guided bone lid in hard mandibular pathosis in term of bone healing.

DETAILED DESCRIPTION:
Mandibular cysts, tumors, and impacted teeth are common pathosis that affect the oral and maxillofacial region, causing bone resorption, swelling, facial asymmetry, infection, and influence quality of life. Such pathosis requires its removal surgically for the preservation of mandibular structure and to avoid complex complications.

Conventional technique for removal of these pathosis requires excessive bone removal with limited accessibility and carries a high possibility of injury to vital structures. On the other hand, the buccal bone lid technique, especially when combined with piezoelectrical devices, demonstrates superiority in preserving vital structures, improving visibility, and enhancing bone healing.

The buccal bone lid acts as a barrier against soft tissue invasion and a reservoir for osteoblasts, that's why it is considered a technique for guided bone regeneration.

Computer-guided surgery and 3d printing guides are essential tools in managing oral and maxillofacial lesion providing patient-specific solutions with high accuracy and predictable outcomes.

A scoping review identified a gap of knowledge regarding the effect of computer-guided surgery in the buccal bone lid technique.

The periosteum is primarily structured by two layers: a superficial outer fibrous layer composed of collagen fibers, elastic fibers, and fibroblasts, and an inner cambium layer rich in fibroblasts, osteoblasts, and a specific type of undifferentiated mesenchymal cells known as periosteal skeletal stem cells (P-SSCs) Shi et al. had reported that P-SSCs have been shown to exhibit pluripotency in vitro, having the ability to differentiate into adipogenic, chondrogenic, and osteogenic lineages, and therefore Inner cambium layer has a great influence on bone remodeling and healing in cases of bone fractures and craniofacial bone injuries Debnath et al. revealed that, unlike bone marrow-derived stem cells (BMSCs), which are involved in endochondral ossification, P-SSCs directly differentiate into osteoblasts via an intramembranous pathway under normal physiological conditions in vivo. However, under pathological conditions, P-SSCs can acquire an endochondral osteogenic capacity after periosteal damage and participate in fracture healing and repair.

The periosteum may retain cell viability if handled properly and stored under appropriate conditions. It can remain viable for less than 1 hour in dry conditions; however, in moist conditions (e.g., saline-soaked gauze), viability may be maintained for up to 2-3 hours. Steiner and Ramp had reported up to 5H preservation in normal saline, Cryopreservation or storage in special preservation media can prolong viability for several days to weeks.

While with full thickness flap elevation, periosteum stripping and elevation from the cortical bone, then repositioned in situ, healing progresses predictably. Within just a few days, early reattachment begins thanks to fibrin deposition and cellular infiltration. By approximately two weeks post-surgery, a newly regenerated periosteal layer is established, complete with osteogenic cells and vascular networks, allowing normal bone-healing activity.

Several studies have examined the biological potential of the periosteum in regenerative contexts. Gamal and Mailhot reported superior clinical and radiographic results using marginal periosteal pedicle grafts (MPP) as guided tissue membranes for treating proximal intrabony defects compared to open flap debridement. Later, Gamal et al. observed coarse-fibered woven bone and cementum-like tissue formation in histological samples 9 months after using MPP.

Ghallab et al. also confirmed that autogenous pedicled periosteal grafts were as effective as bioresorbable collagen membranes in improving clinical and radiographic outcomes for intra-bony periodontal defects Puisys et al. Clinically evaluated connective tissue grafts from the tuberosity for increasing soft tissue thickness and keratinization in edentulous mandibles. They found that keratinization of non-keratinized mucosa was more pronounced in partial-thickness flap groups.

Fickl et al. examined the effect of flap thickness on bone loss and reported that partial-thickness flaps, although not preventing bone loss, resulted in less bone loss compared to full-thickness flaps Mounir et al. Similarly had reported reduced marginal bone loss in maxillary ridge-splitting procedures using split-thickness flaps compared to full-thickness flaps.

To our knowledge, the technique of using a split-thickness flap with a guided bone lid approach for managing mandibular pathosis is novel. Based on the periosteum's unique role in osteogenesis and regeneration, its preservation by keeping it attached to the bone lid during temporary removal may enhance healing. This technique requires investigation, particularly in the context of avoiding periosteum stripping and maintaining lid vascularity

ELIGIBILITY:
Inclusion criteria:

* No sex predilection.
* Age: 18 to 40
* mandibular intra-bony hard pathosis with a diameter ≥1cm with a buccal cortex thickness ≥1mm

Exclusion criteria:

* Systemic or local disease/ condition that could affect bone healing
* Diabetics
* patients on systemic corticosteroid
* chemotherapy
* radiotherapy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
• bone defect filling | 6 months
  bone healing will be measured with Cone beam CT

SECONDARY OUTCOMES:
• Intra-operative time | intra operative time needed for both techniques
• Pain | first , third . 7th day post operative
  • Pain will be measured by visual analogue scale VAS with 0 indicating no pain and 10 indicating the most severe pain. Patients will be asked to score the pain based on severity on the first, third, and seventh days
• Accuracy of transfer of the cutting guide | immediate post operative using the post operative CBCT
  • Guide/osteotomy accuracy in millimeters, by superimposing the preoperative virtual guide outline based on the preoperative Cone Beam Computer Tomography (CBCT) and the immediate post operative actual osteotomy lines on postoperative CBCT

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sivolella S, Brunello G, Panda S, Schiavon L, Khoury F, Del Fabbro M. The Bone Lid Technique in Oral and Maxillofacial Surgery: A Scoping Review. J Clin Med. 2022 Jun 24;11(13):3667. doi: 10.3390/jcm11133667. PMID 35806950
- [Background] Mounir M, Beheiri G, El-Beialy W. Assessment of marginal bone loss using full thickness versus partial thickness flaps for alveolar ridge splitting and immediate implant placement in the anterior maxilla. Int J Oral Maxillofac Surg. 2014 Nov;43(11):1373-80. doi: 10.1016/j.ijom.2014.05.021. Epub 2014 Jun 25. PMID 24973295
- [Background] Khoury F, Hanser T. Mandibular bone block harvesting from the retromolar region: a 10-year prospective clinical study. Int J Oral Maxillofac Implants. 2015 May-Jun;30(3):688-97. doi: 10.11607/jomi.4117. PMID 26009921
- [Background] Gamal AY, Mailhot JM. A novel marginal periosteal pedicle graft as an autogenous guided tissue membrane for the treatment of intrabony periodontal defects. J Int Acad Periodontol. 2008 Oct;10(4):106-17. PMID 19055224
- [Background] Fickl S, Kebschull M, Schupbach P, Zuhr O, Schlagenhauf U, Hurzeler MB. Bone loss after full-thickness and partial-thickness flap elevation. J Clin Periodontol. 2011 Feb;38(2):157-62. doi: 10.1111/j.1600-051X.2010.01658.x. Epub 2010 Nov 30. PMID 21118288
- [Background] Degerliyurt K, Akar V, Denizci S, Yucel E. Bone lid technique with piezosurgery to preserve inferior alveolar nerve. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Dec;108(6):e1-5. doi: 10.1016/j.tripleo.2009.08.006. PMID 19913713
- [Background] Straubinger RM, Papahadjopoulos D. Liposomes as carriers for intracellular delivery of nucleic acids. Methods Enzymol. 1983;101:512-27. doi: 10.1016/0076-6879(83)01035-6. No abstract available. PMID 6193396
- [Background] Postawa B. [Evaluation of HIV infection progression in patients treated at the Infectious Diseases Clinic of the Jagiellonian University in Cracow in the years 1989-1993]. Folia Med Cracov. 1996;37(1-2):29-47. Polish. PMID 9312524